CLINICAL TRIAL: NCT02837926
Title: Work Package 4: HPV Vaccination of Women in Screening Ages
Brief Title: Comparing Health Services Interventions for the Prevention of HPV-related Cancer
Acronym: CoheaHr-WP4
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: CHU de Reims (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: PO15019
Record Dates: First submitted 2016-07-13; First posted 2016-07-20 (Estimated); Last update posted 2019-04-10 (Actual); Status verified 2019-04

CONDITIONS: Cervical Cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Surveys and Questionnaires; Human Papillomavirus Recombinant Vaccine Quadrivalent, Types 6, 11, 16, 18; human papillomavirus vaccine, L1 type 16, 18

ARMS (1):
- women attending for cervical cancer screening (Experimental)
  Interventions: Other: questionnaire; Biological: Gardasil vaccine; Biological: Cervarix®

INTERVENTIONS:
Other: questionnaire
Biological: Gardasil vaccine
Biological: Cervarix®

SUMMARY:
The study aims to identify global and local determinants of HPV vaccine acceptability, HPV vaccine uptake and compliance as well as identify logistics and programmatic issues in each country to offer the HPV vaccine, as a potential cervical cancer prevention strategy, to mid-aged women attending screening.

DETAILED DESCRIPTION:
3000 women aged within the age range of 25-45 years old will be recruited; 250-300 women per country. These women will be identified by means of screening registry lists or screening clinical visits. Eligible women will receive a study questionnaire on the HPV vaccine. Additionally, and independently of participating in the study questionnaire, those who accept will get 3 HPV vaccine doses. Depending on country preferences, either Cervarix® (Glaxosmithkline Biologicals, S.A.) at month 0, 1 and 6 or Gardasil® (Sanofi Pasteur MSD SNC) at month 0, 2 and 6, will be administered.

Safety data and HPV vaccine compliance will be assessed.

A sub study in Spain will also analyze acceptability of HPV vaccination in a sample of women aged 35-40 yrs identified as poor screening attenders.

Two independent informed consent forms will be provided; one for the study questionnaire participation and another for HPV vaccine administration.

ELIGIBILITY:
Inclusion Criteria:

* women within the age range of 25-45
* attending cervical cancer screening

Exclusion Criteria:

* previous history of HPV vaccine administration

Ages: 25 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 63 (Actual)
Dates: Start 2016-05; Primary Completion 2017-12 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
number of vaccinated patients | up to 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Reims, Reims, France